CLINICAL TRIAL: NCT02711553
Title: Randomized, Double-Blind, Phase 2 Study of Ramucirumab or Merestinib or Placebo Plus Cisplatin and Gemcitabine as First-Line Treatment in Patients With Advanced or Metastatic Biliary Tract Cancer
Brief Title: A Study of Ramucirumab (LY3009806) or Merestinib (LY2801653) in Advanced or Metastatic Biliary Tract Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16329; I3O-MC-JSBF (Other: Eli Lilly and Company); 2015-004699-31 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Cancer; Metastatic Cancer; Advanced Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasm Metastasis | interventions — Ramucirumab; merestinib; Cisplatin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (Experimental): Participants received 8 mg/kg ramucirumab plus 25 mg/square meter (mg/m²) cisplatin and 1000 mg/m² gemcitabine intravenously (IV) on days 1 and 8, every 21 days (1 cycle). Participants may continue on study drug for up to 8 cycles (for cisplatin and gemcitabine therapy) or until disease progression, unacceptable toxicity, or other withdrawal criterion is met (for ramucirumab therapy).
  Interventions: Drug: Ramucirumab; Drug: Cisplatin; Drug: Gemcitabine
- Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (Placebo Comparator): Participants received placebo (indistinguishable and equivalent volume to ramucirumab) plus 25 mg/m² cisplatin and 1000 mg/m² gemcitabine IV on days 1 and 8, every 21 days (1 cycle). Participants may continue on study drug for up to 8 cycles (for cisplatin and gemcitabine therapy) or until disease progression, unacceptable toxicity, or other withdrawal criterion is met (for placebo therapy).
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Placebo IV
- 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (Experimental): Participants received 80 mg merestinib orally each day, plus 25 mg/m² cisplatin and 1000 mg/m² gemcitabine IV on Days 1 and 8, every 21 days (1 cycle). Participants may continue on study drug for up to 8 cycles (for cisplatin and gemcitabine therapy) or until disease progression, unacceptable toxicity, or other withdrawal criterion is met (for merestinib therapy).
  Interventions: Drug: Merestinib; Drug: Cisplatin; Drug: Gemcitabine
- Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (Placebo Comparator): Participants received placebo (indistinguishable to merestinib) orally each day, plus 25 mg/m² cisplatin and 1000 mg/m² gemcitabine IV on Days 1 and 8, every 21 days. Participants may continue on study drug for up to 8 cycles (for cisplatin and gemcitabine therapy) or until disease progression, unacceptable toxicity, or other withdrawal criterion is met (for placebo therapy).
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Placebo Oral

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Drug: Merestinib — Administered orally
  Other Names: LY2801653
  Arms: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Drug: Cisplatin — Administered IV
Drug: Gemcitabine — Administered IV
  Other Names: LY188011
Drug: Placebo Oral — Administered orally
  Arms: Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Drug: Placebo IV — Administered IV
  Arms: Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of ramucirumab or merestinib or placebo plus cisplatin and gemcitabine in participants with advanced or metastatic biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have a histologically or cytologically confirmed diagnosis of non-resectable, recurrent, or metastatic biliary tract adenocarcinoma (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer, or Ampulla of Vater) .
* Have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
* Have adequate biliary drainage.
* Have adequate organ function.
* Males and females are sterile, postmenopausal, or compliant with a highly effective contraceptive method.
* Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose.
* Are willing to provide blood/serum/plasma and tumor tissue samples for research purposes. Submission of blood/serum/plasma and tumor tissue samples is mandatory for participation in this study, unless restricted per local regulations.

Exclusion Criteria:

* Previous systemic therapy for locally advanced or metastatic disease is not allowed.
* Have a history of or have current hepatic encephalopathy of any grade, or ascites of Grade >1, or cirrhosis with Child-Pugh Stage B or higher.
* Have ongoing or recent (≤6 months) hepatorenal syndrome.
* Have had a major surgical procedure or significant traumatic injury including nonhealing wound, peptic ulcer, or bone fracture ≤28 days prior to randomization.
* Anticipate having a major surgical procedure during the course of the study.
* Has documented brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression.
* Within 6 months prior to randomization, have had any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack.
* Have an uncontrolled arterial hypertension with systolic blood pressure ≥150 or diastolic blood pressure ≥90 millimeters of mercury (mm Hg) despite standard medical management.
* Have a previous malignancy within 5 years of study entry or a concurrent malignancy.
* Have a history of gastrointestinal perforation and/or fistulae within 6 months prior to randomization.
* Have a known allergy or hypersensitivity reaction to any of the treatment components.
* Have a history of uncontrolled hereditary or acquired thrombotic disorder.
* Have uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain.
* Have mixed hepatocellular biliary tract cancer histology.
* Have a corrected QT interval >470 milliseconds as calculated by the Fridericia equation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (81):
- United States (12):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida School of Medicine, Gainesville, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University Medical School, City of Saint Peters, Missouri
  - Washington University Medical School, Creve Coeur, Missouri
  - Washington University Medical School, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Florida Cancer Specialists, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Argentina (8):
  - Alexander Fleming, CABA, BS
  - Hospital de Gastroenterologia Udaondo, Capital Federal, Buenos Aires
  - Fundacion Ars Medica, San Salvador de Jujuy, Jujuy Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Fundacion Favaloro, Ciudad de Buenos Aires
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
  - Centro Polivalente de Asistencia e Inv. Clinica CER-San Juan, San Juan
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
- Austria (3):
  - Landesklinikum Wr. Neustadt, Wiener Neustadt, Lower Austria
  - Universitätsklinikum Salzburg, Salzburg
  - KH der Barmherzigen Brüder Wien, Vienna
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels, Brussels Capital
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice v Motole, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus Sygehus, Aarhus C
  - Odense Universitetshospital, Odense C
- France (7):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - CHU de Bordeaux Hop St ANDRE, Bordeaux, Gironde
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - Hôpital C. HURIEZ, Lille
  - CHRU de Montpellier-Hopital St Eloi, Montpellier
  - Centre Antoine-Lacassagne, Nice
  - Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Medizinische Hochschule Hanover, Hanover, Lower Saxony
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont Onkologiai Tanszek, Debrecen, Hajdú-Bihar
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
- Mexico (2):
  - Arke Estudios Clinicos S.A. de C.V., Mexico City, Mexico City
  - Centro de Alta Especialidad Reumatologia Inv del Potosi SC, San Luis Potosí City
- Russia (4):
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg, Sankt-Peterburg
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Blokhin Cancer Research Center, Moscow
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
- South Korea (4):
  - Asan Medical Center, Seoul, Korea
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínico Universitario de Valencia, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico de San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (2):
  - Skåne universitetssjukhus, Malmo
  - Karolinska Universitetssjukhuset i Solna, Stockholm
- Taiwan (5):
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- Turkey (Türkiye) (5):
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Hacettepe University Faculty of Medicine, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Trakya University, Edirne
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi Yerleskesi, Istanbul
- United Kingdom (5):
  - University College Hospital - London, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Hammersmith Hospital, Acton, London
  - The Clatterbridge Cancer Centre, Bebbington, Merseyside
  - Royal Marsden Hospital, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Valle JW, Vogel A, Denlinger CS, He AR, Bai LY, Orlova R, Van Cutsem E, Adeva J, Chen LT, Obermannova R, Ettrich TJ, Chen JS, Wasan H, Girvan AC, Zhang W, Liu J, Tang C, Ebert PJ, Aggarwal A, McNeely SC, Moser BA, Oliveira JM, Carlesi R, Walgren RA, Oh DY. Addition of ramucirumab or merestinib to standard first-line chemotherapy for locally advanced or metastatic biliary tract cancer: a randomised, double-blind, multicentre, phase 2 study. Lancet Oncol. 2021 Oct;22(10):1468-1482. doi: 10.1016/S1470-2045(21)00409-5. PMID 34592180
- See also: A Study of Ramucirumab (LY3009806) or Merestinib (LY2801653) in Advanced or Metastatic Biliary Tract Cancer — https://trials.lillytrialguide.com/en-US/trial/3MKeCKU0hiwqg4gsAMgAEs

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Participant Flow, participants who completed were those who died due to any cause or were alive and on study at conclusion but off treatment.
Period: Overall Study
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Started | 106 | 52 | 102 | 49
Received at Least 1 Dose of Study Drug | 104 | 52 | 102 | 48
Completed | 100 | 47 | 92 | 45
Not Completed | 6 | 5 | 10 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 3 | 6 | 3
Not completed — On Study Treatment at Study Conclusion | 1 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine: Participants received 8 mg/kg ramucirumab plus 25 mg/m² cisplatin and 1000 mg/m² gemcitabine IV on days 1 and 8, every 21 days (1 cycle). Participants may continue on study drug for up to 8 cycles (for cisplatin and gemcitabine therapy) or until disease progression, unacceptable toxicity, or other withdrawal criterion is met (for ramucirumab therapy).
- Total: Total of all reporting groups
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Total
Number analyzed (Participants) | 106 | 52 | 102 | 49 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.49 (9.76) | 57.06 (11.67) | 60.95 (9.14) | 62.00 (9.14) | 61.33 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized participants and all randomized participants who received at least 1 dose of study drug to align gender specific adverse event numbers.
  Participants
    All randomized participants: Female | 60 | 26 | 54 | 22 | 162
    All randomized participants: Male | 46 | 26 | 48 | 27 | 147
    All randomized participants who received at least 1 dose of study drug: number analyzed (Participants) | 104 | 52 | 102 | 48 | 306
    All randomized participants who received at least 1 dose of study drug: Female | 59 | 26 | 54 | 21 | 160
    All randomized participants who received at least 1 dose of study drug: Male | 45 | 26 | 48 | 27 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 106 | 52 | 102 | 49 | 309
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 20 | 11 | 26 | 9 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  White | 78 | 35 | 70 | 38 | 221
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 4 | 1 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 11 | 3 | 8 | 3 | 25
  Hungary | 5 | 7 | 4 | 1 | 17
  United States | 12 | 3 | 6 | 4 | 25
  Czechia | 2 | 2 | 5 | 2 | 11
  United Kingdom | 4 | 2 | 5 | 3 | 14
  Russia | 9 | 2 | 4 | 6 | 21
  Spain | 8 | 3 | 10 | 1 | 22
  Austria | 3 | 2 | 1 | 0 | 6
  South Korea | 8 | 6 | 12 | 4 | 30
  Sweden | 1 | 0 | 3 | 2 | 6
  Turkey | 6 | 7 | 7 | 3 | 23
  Belgium | 6 | 1 | 3 | 4 | 14
  Taiwan | 9 | 5 | 13 | 4 | 31
  Denmark | 1 | 1 | 3 | 1 | 6
  Mexico | 4 | 0 | 3 | 0 | 7
  Australia | 6 | 2 | 2 | 4 | 14
  France | 8 | 5 | 5 | 2 | 20
  Germany | 3 | 1 | 8 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS time was measured from the date of randomization until the first radiographic documentation of progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Randomization to Progressive Disease or Death from Any Cause (Up To 20 Months)
Population: All randomized participants. Censored participants: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine = 29; 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine = 34; Pooled Placebo = 25. Pooling is done in the placebo arm (Pooled Placebo) from both arms (Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine and Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine) for analysis purpose and combined as pre-specified in protocol.
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Pooled Placebo: Participants received placebo IV and placebo oral (indistinguishable and equivalent volume to ramucirumab and merestinib) plus 25 mg/m² cisplatin and 1000 mg/m² gemcitabine IV on days 1 and 8, every 21 days (1 cycle). Participants may continue on study drug for up to 8 cycles (for cisplatin and gemcitabine therapy) or until disease progression, unacceptable toxicity, or other withdrawal criterion is met (for placebo therapy).
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 106 | 102 | 101
Months | 6.47 [3.68 to 8.51] | 6.97 [4.34 to 9.79] | 6.64 [4.11 to 9.72]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.4821, Log Rank — p-value is 2-sided; Stratified by geographical region, pathological diagnosis, metastatic disease; Hazard Ratio (HR) = 1.123, 80% CI 2-sided [0.904 to 1.395] — Stratified by geographical region, pathological diagnosis, metastatic disease
Statistical Analysis 2: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.6417, Log Rank — p-value is 2-sided; Stratified by geographical region, pathological diagnosis, metastatic disease; Hazard Ratio (HR) = 0.920, 80% CI 2-sided [0.734 to 1.153] — Stratified by geographical region, pathological diagnosis, metastatic disease

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from from randomization to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: Randomization to Date of Death from Any Cause (Up To 48 Months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 106 | 102 | 101
Months | 10.45 [8.48 to 11.76] | 14.03 [11.96 to 16.36] | 13.04 [11.40 to 15.31]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.0870, Log Rank; Stratified by geographical region, pathological diagnosis, metastatic disease; Hazard Ratio (HR) = 1.336, 95% CI 2-sided [0.959 to 1.862] — Stratified by geographical region, pathological diagnosis, metastatic disease
Statistical Analysis 2: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.7599, Log Rank; Stratified by geographical region, pathological diagnosis, metastatic disease; Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.669 to 1.342] — Stratified by geographical region, pathological diagnosis, metastatic disease

3. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR): Objective Response Rate (ORR)
Description: ORR was the number of participants who achieve a best overall response of CR or PR divided by the total number of participants randomized to the corresponding treatment arm as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Disease Progression (Up To 30 Months)
Population: All randomized participants. Pooling is done in the placebo arm (Pooled Placebo) from both arms (Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine and Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine) for analysis purpose and combined as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 106 | 102 | 101
Percentage of participants | 31.1 [22.3 to 39.9] | 19.6 [11.9 to 27.3] | 32.7 [23.5 to 41.8]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.878, Exact Cochran-Mantel-Haenszel; Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.9] — Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease
Statistical Analysis 2: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.023, Exact Cochran-Mantel-Haenszel; Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.2 to 0.9] — Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease

4. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD): Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was the number of participants who achieve a best overall response of CR, PR, or SD divided by the total number of participants randomized to the corresponding treatment arm as per RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Disease Progression (Up To 30 Months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 106 | 102 | 101
Percentage of participants | 81.1 [73.7 to 88.6] | 83.3 [76.1 to 90.6] | 78.2 [70.2 to 86.3]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.680, Exact Cochran-Mantel-Haenszel; Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.6 to 2.4] — Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease
Statistical Analysis 2: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; Test type: Superiority; p = 0.499, Exact Cochran-Mantel-Haenszel; Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.6 to 2.6] — Stratified by randomization strata Geographical Region, Pathological Diagnosis, Metastatic Disease

5. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Description: PK was determined by the minimum observed plasma concentration (Cmin). 1 Cycle (C) = 21 days (D).
Time Frame: C1 D8, C2 D1, C3 D1, C4 D1,C5 D1,C7 D1, C9 D1 and C13 D1: Within 3 days Prior to Infusion(PTI)
Population: All participants who received at least one dose of study drug and had evaluable PK data. As per protocol, Cmin of merestinib was not measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (µg/mL)
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Number analyzed (Participants) | 86
Microgram per milliliter (µg/mL)
  Cycle 1 Day 8 (Week 1) | 46.2 (32)
  Cycle 2 Day 1 (Week 3): number analyzed (Participants) | 74
  Cycle 2 Day 1 (Week 3) | 38.1 (42)
  Cycle 3 Day 1 (Week 6): number analyzed (Participants) | 53
  Cycle 3 Day 1 (Week 6) | 54.1 (43)
  Cycle 4 Day 1 (Week 9): number analyzed (Participants) | 48
  Cycle 4 Day 1 (Week 9) | 77.3 (50)
  Cycle 5 Day 1 (Week 12): number analyzed (Participants) | 32
  Cycle 5 Day 1 (Week 12) | 82.9 (35)
  Cycle 7 Day 1 (Week 18): number analyzed (Participants) | 19
  Cycle 7 Day 1 (Week 18) | 85.6 (39)
  Cycle 9 Day 1 (Week 24): number analyzed (Participants) | 9
  Cycle 9 Day 1 (Week 24) | 82.7 (35)
  Cycle 13 Day 1 (Week 36): number analyzed (Participants) | 7
  Cycle 13 Day 1 (Week 36) | 97.7 (23)

6. Secondary Outcome: PK: Plasma Concentration of Merestinib
Description: PK was presented through graphical overlay comparison versus historic data. No numerical summary of data was intended or produced.
Time Frame: C1 D8; C2 D1; C4 D1; C6 D1; C8 D1; C2 D8; C4 D8; C6 D8; C8 D8: Morning
Population: Zero participants were analyzed as no data collected for summary analysis.
Arm/Group | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Ramucirumab Antibodies
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies (ADA) was summarized by treatment group.
Time Frame: Predose Cycle 1 Day 1 through Follow Up (Up To 48 Months)
Population: All randomized participants who received at least 1 dose of study drug with both baseline and at least one post baseline ADA assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
Number analyzed (Participants) | 74 | 37
Participants | 3 | 0

8. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy Hepatobiliary Questionnaire (FACT-Hep)
Description: FACT-Hep consists of 45 items in five subscales (1) physical well-being (PWB) score rage 0 -28; (2) social well-being (SWB) score range 0-28; (3) emotional well-being (EWB) score range 0-24; (4) functional well-being (FWB) score range 0-28; and (5) the hepatobiliary cancer subscale (HCS) Score range 0-72. The Trial Outcomes Index (TOI) is the sum of the PWB, FWB and Hep subscales with a scores range of 0 to 128. The Total FACT-Hep score was the sum of all questions with a scores range of 0 to 180.Total FACT-G score was the sum of the 27 questions in the PWB, SFWB, EWB and FWB with a scores range of 0 to 108. The FACT-Hep Symptoms Index with 8 key questions and scores range of 0 to 32 from the Hep Subscale. Higher score in sub-score or total score indicates better QOL and better health state. Participants were classified as "Improved" if they had positive change from baseline, "Worsened" if they had negative change from baseline, and "Stable" otherwise.
Time Frame: Baseline, Follow Up (Up To 48 Months)
Population: All randomized participants who received at least 1 dose of study drug with baseline and one post-baseline FACT-Hep Questionnaire.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 97 | 95 | 95
Units on a Scale
  PWB | -2.75 (0.43) | -2.88 (0.43) | -1.65 (0.42)
  SWB | -0.26 (0.36) | 0.22 (0.36) | 0.56 (0.36)
  EWB | 0.23 (0.31) | 0.64 (0.32) | 0.93 (0.31)
  FWB | -2.40 (0.44) | -1.34 (0.44) | -0.75 (0.44)
  HCS | -3.62 (0.63) | -2.32 (0.64) | -0.68 (0.63)
  FACT-Hep | -1.11 (0.37) | -0.74 (0.37) | -0.09 (0.37)
  TOI | -8.68 (1.31) | -6.43 (1.32) | -3.01 (1.30)
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; PWB; Test type: Superiority; p = 0.069, MMRM Model — p-values are from Type 3 sums of squares mixed model repeated measures (MMRM) Model; Least Squares (LS) Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -1.10, 95% CI 2-sided [-2.28 to 0.09], Standard Error of Mean 0.60
Statistical Analysis 2: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; PWB; Test type: Superiority; p = 0.042, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -1.23, 95% CI 2-sided [-2.42 to -0.04], Standard Error of Mean 0.60
Statistical Analysis 3: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine; SWB; Test type: Superiority; p = 0.112, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -0.82, 95% CI 2-sided [-1.83 to 0.19], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; SWB; Test type: Superiority; p = 0.505, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -0.34, 95% CI 2-sided [-1.35 to 0.67], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; EWB; Test type: Superiority; p = 0.116, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -0.70, 95% CI 2-sided [-1.56 to 0.17], Standard Error of Mean 0.44
Statistical Analysis 6: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; EWB; Test type: Superiority; p = 0.521, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -0.29, 95% CI 2-sided [-1.16 to 0.59], Standard Error of Mean 0.45
Statistical Analysis 7: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; FWB; Test type: Superiority; p = 0.008, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -1.66, 95% CI 2-sided [-2.87 to -0.44], Standard Error of Mean 0.62
Statistical Analysis 8: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; FWB; Test type: Superiority; p = 0.335, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -0.60, 95% CI 2-sided [-1.82 to 0.62], Standard Error of Mean 0.62
Statistical Analysis 9: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; HCS; Test type: Superiority; p = 0.001, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -2.93, 95% CI 2-sided [-4.69 to -1.18], Standard Error of Mean 0.89
Statistical Analysis 10: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; HCS; Test type: Superiority; p = 0.068, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -1.64, 95% CI 2-sided [-3.40 to 0.12], Standard Error of Mean 0.89
Statistical Analysis 11: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; FACT-Hep; Test type: Superiority; p = 0.051, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -1.02, 95% CI 2-sided [-2.04 to 0.00], Standard Error of Mean 0.52
Statistical Analysis 12: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; FACT-Hep; Test type: Superiority; p = 0.212, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -0.65, 95% CI 2-sided [-1.68 to 0.38], Standard Error of Mean 0.52
Statistical Analysis 13: Comparison: 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; TOI; Test type: Superiority; p = 0.002, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -5.67, 95% CI 2-sided [-9.30 to -2.04], Standard Error of Mean 1.84
Statistical Analysis 14: Comparison: 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine vs Pooled Placebo; TOI; Test type: Superiority; p = 0.066, MMRM Model — p-values are from type 3 sums of squares MMRM model; LS Mean value was adjusted for treatment, visit, baseline, treatment*visit and baseline*visit; LS Mean Difference = -3.42, 95% CI 2-sided [-7.07 to 0.22], Standard Error of Mean 1.85

9. Secondary Outcome: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Score
Description: EQ-5D-5L is a 2-part questionnaire that assesses general health status for 'today'. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using country-specific algorithms, with scores ranging from less than 0 (where zero is a health state equivalent to death; negative values are valued as worse than dead) to 1 (perfect health). Index values were calculated using the US algorithm (-0.109 to 1). A higher score indicates better health state.
Time Frame: Baseline, Follow Up (Up To 48 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 5L data.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 45 | 42 | 40
Units on a Scale | 0.61 (0.31) | 0.63 (0.29) | 0.66 (0.27)

10. Secondary Outcome: Change From Baseline in Participant-Reported EQ-5D-5L Visual Analog Scale (VAS) Score
Description: EQ-5D-5L is a 2-part questionnaire that assesses general health status 'today'. The second part is assessed using a VAS on which the patient rates their perceived health state, ranging from 0 millimeter (the worst health you can imagine) to 100 millimeter (the best health you can imagine).
Time Frame: Baseline, Follow Up (Up To 48 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 5L data.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Pooled Placebo
Number analyzed (Participants) | 45 | 42 | 40
millimeter (mm) | 66.44 (22.8) | 66.57 (21.73) | 69.08 (20.03)

ADVERSE EVENTS:
Time Frame: Randomization Up To 48 Months
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine | Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine
All-Cause Mortality (participants affected / at risk) | 84/104 | 34/52 | 71/102 | 38/48
Serious Adverse Events (participants affected / at risk) | 53/104 | 25/52 | 56/102 | 23/48
Other Adverse Events (participants affected / at risk) | 102/104 | 49/52 | 100/102 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=104) | Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=52) | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=102) | Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=48)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 5 (5) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 3 (3) | 2 (2) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5) | 0 (0)
Anastomotic ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 4 (5) | 1 (1)
Catheter site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (9) | 1 (1) | 4 (5) | 2 (4)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 5 (7) | 0 (0) | 2 (2) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 3 (6) | 1 (1) | 2 (3) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Meningitis meningococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 1 (2) | 4 (6) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg Ramucirumab + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=104) | Placebo IV + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=52) | 80 mg Merestinib + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=102) | Placebo Oral + 25 mg/m² Cisplatin + 1000 mg/m² Gemcitabine (N=48)
Anemia (Blood and lymphatic system disorders) | 52 (94) | 22 (39) | 40 (80) | 24 (33)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 20 (45) | 9 (23) | 20 (46) | 4 (15)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (3) | 2 (3) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 63 (160) | 24 (63) | 52 (122) | 19 (60)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 56 (120) | 15 (31) | 42 (80) | 15 (33)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 4 (7) | 0 (0) | 3 (5) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 10 (13) | 2 (2) | 14 (15) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 39 (54) | 13 (27) | 33 (47) | 15 (26)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 13 (13) | 2 (2) | 10 (11) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 33 (49) | 14 (23) | 36 (59) | 13 (16)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 34 (50) | 9 (10) | 29 (36) | 7 (13)
Dry mouth (Gastrointestinal disorders) | 5 (11) | 1 (1) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (8) | 2 (6) | 4 (5) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (5) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 52 (92) | 21 (39) | 58 (97) | 15 (24)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 11 (15) | 5 (7) | 4 (6) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 34 (130) | 12 (18) | 34 (93) | 12 (26)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 8 (18) | 1 (1) | 5 (8) | 2 (2)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 5 (7) | 1 (1) | 7 (10) | 2 (2)
Fatigue (General disorders) | 61 (94) | 17 (22) | 53 (90) | 22 (34)
Gait disturbance (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (3) | 2 (2) | 3 (4) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (2)
Oedema (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 33 (46) | 7 (10) | 18 (22) | 6 (9)
Pain (General disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Pyrexia (General disorders) | 25 (46) | 6 (12) | 26 (52) | 9 (11)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 3 (6) | 1 (1) | 3 (3) | 4 (4)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hepatic infarction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Portal vein stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 4 (4) | 1 (2) | 3 (3) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 2 (2) | 3 (4) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 4 (5) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 4 (7) | 7 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 11 (17) | 2 (2) | 8 (9) | 2 (4)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (18) | 6 (9) | 32 (55) | 7 (11)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 14 (19) | 9 (11) | 26 (38) | 8 (10)
Bacterial test (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 9 (12) | 8 (12) | 10 (13) | 3 (3)
Blood bilirubin increased (Investigations) | 15 (16) | 4 (4) | 11 (14) | 5 (5)
Blood creatinine increased (Investigations) | 10 (16) | 4 (4) | 11 (19) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Computerised tomogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eastern cooperative oncology group performance status worsened (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 6 (8) | 6 (7) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Paracentesis (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Urine output decreased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Wall motion score index abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 16 (18) | 3 (3) | 14 (15) | 7 (7)
Weight increased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 39 (47) | 14 (14) | 26 (41) | 14 (17)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (12) | 3 (3) | 3 (4) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1) | 5 (5) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (14) | 6 (7) | 11 (15) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 8 (9) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (15) | 3 (3) | 9 (12) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 (32) | 8 (11) | 10 (11) | 7 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (17) | 4 (5) | 4 (7) | 4 (5)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 4 (7) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 6 (6) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (19) | 8 (9) | 9 (10) | 7 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (4) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 3 (4) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (5) | 5 (5) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (4) | 7 (7) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allodynia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 10 (17) | 4 (5) | 12 (14) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 12 (15) | 1 (1) | 8 (10) | 4 (4)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (21) | 8 (12) | 14 (18) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 16 (21) | 5 (7) | 23 (32) | 5 (5)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 7 (10) | 0 (0) | 2 (2) | 3 (3)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (6) | 2 (2) | 0 (0) | 2 (6)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 3 (4) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 5 (6) | 9 (9) | 5 (5)
Pressure of speech (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 3 (3) | 3 (3) | 0 (0)
Chromaturia (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 13 (18) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (4) | 1 (1) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 3 (4) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 0 (0) | 8 (9) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 7 (7) | 8 (11) | 10 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (27) | 2 (2) | 2 (2) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 7 (7) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13) | 3 (3) | 14 (14) | 8 (8)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 2 (2) | 9 (9) | 7 (7)
Purpura (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (12) | 1 (1) | 7 (19) | 3 (3)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Respite care (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Cholangiostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Embolism arterial (Vascular disorders) | 2 (3) | 1 (1) | 4 (4) | 0 (0)
Embolism venous (Vascular disorders) | 3 (3) | 1 (1) | 6 (6) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 32 (53) | 2 (2) | 6 (11) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Lymphoedema (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement is maximum of 10 years restriction on the PI that the sponsor can review results communications prior to public release and can embargo communications regarding trial results. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02711553/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02711553/SAP_001.pdf